CLINICAL TRIAL: NCT04412460
Title: Echocardiography in Patients With Covid-19 Undergoing Intensive Care Therapy
Brief Title: Echocardiography in Patients With Covid-19
Status: Withdrawn | Type: Observational
Why Stopped: Not feasible.
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: CovidEcho
Record Dates: First submitted 2020-05-20; First posted 2020-06-02 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2020-05

CONDITIONS: COVID; ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective observational study of patients treated due to Covid-19 disease. Observation and analysis of echocardiographic studies performed in the intensive care setting.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Covid-19 disease
* invasive Ventilation

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults admitted for ICU therapy due to severe Covid-19
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
ICU Mortality | up to 90 days

SECONDARY OUTCOMES:
ICU length-of stay | up to 90 days
ICU ventilator free days | up to 90 days
Hospital length-of-stay | up to 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tubingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No